CLINICAL TRIAL: NCT04682912
Title: ABO-Rh Blood Types and COVID-19 Infection in Children: Is There a Link?
Brief Title: Blood Types in Children With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mersin Training and Research Hospital (Other Government)
Collaborators: Mersin University (Other); Dicle University (Other); Bezmialem Vakif University (Other); Uludag University (Other)
Responsible Party: Principal Investigator, Ali Özdemir, Assoc Prof Ali Özdemir, Mersin Training and Research Hospital
Other Study IDs: MersinTRH
Record Dates: First submitted 2020-12-22; First posted 2020-12-24 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; ABO blood group; infection risk
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is speculated that in adult patients with COVID-19 blood type A is associated with the worst outcome, while blood type O is associated with mild symptoms.To our knowledge, there has been no such a study investigated ABO and Rhesus (Rh) blood group types in children with COVID-19 infection yet. Therefore, the study aimed to examine if such a correlation exists in children infected with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* The study period consisted between March 2020 and December 2020
* Children with a documented positive COVID-19 nasal smear real-time reverse-transcriptase polymerase chain reaction (PCR) assay were included.

Exclusion Criteria:

* Patients who had a past medical history of any chronic illness (related to respiratory, cardiology, immunology, neurology, metabolic, etc) were excluded.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A retrospective multicenter trial in five major hospitals in Turkey to determine whether ABO and Rh blood types carry any risk/beneficial factor among children with COVID-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Patient medical files | 1 month
  ABO blood type distribution will be different in COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Ali̇ Özdemi̇r, MD, Principal Investigator — Mersi̇n Şehi̇r Eği̇ti̇m Ve Araşti̇rma Hastanesi̇; Ali̇ Özdemi̇r, Principal Investigator — Mersi̇n Şehi̇r Eği̇ti̇m Ve Araşti̇rma Hastanesi̇
Locations (1):
- Mersin City Training & Research Hospital, Mersi̇n, Turkey (Türkiye)